CLINICAL TRIAL: NCT03620253
Title: Does Modafinil Have Pro-cognitive Effects in Those With Residual Cognitive Impairment Despite Remitted Depression?
Brief Title: Modafinil's Effects on Cognition in Remitted MDD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Principal Investigator left study site
Sponsor: Unity Health Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); The Canadian Biomarker Integration Network in Depression (Unknown)
Responsible Party: Principal Investigator, Shane McInerney, Staff Psychiatrist, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOCOG-01
Record Dates: First submitted 2018-07-27; First posted 2018-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder; Cognitive Impairment
Keywords: modafinil; remitted depression; cognition
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction | interventions — Modafinil

STUDY DESIGN:
Intervention Model Description: 50 Participants (aged 18-55) who are experiencing cognitive deficits (measured as Neurocognitive Index >1 standard deviation below the mean) despite remission from depression (Montgomery-Asberg Rating Scale for Depression (MADRAS) score <7) will be eligible to receive modafinil (100-200mg daily) or two identical placebo capsules each morning for a period of 8 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 25 participants will be randomly assigned to the modafinil treatment group, and 25 to the placebo group. The drug/placebo will be randomized and dispensed by the research pharmacy at St. Michael's Hospital. A research technician who is blind to the study will prepare the capsules and break the blind at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modafinil (Experimental): Participants will be administered 100 mg modafinil tablets, that will be over-encapsulated, for one week. If the drug is well tolerated, the dosage will be increased to 200 mg for the remaining 7 weeks of the study. Capsules are taken daily in the morning.
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Participants will be administered 100 mg placebo capsule. This capsule will have all the same ingredients as the modafinil tablets, minus the active ingredient. After 1 week, participants' dosage will be increased to 200 mg for the remaining 7 weeks of the study. Capsules are taken daily in the morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — Participants randomized to the modafinil group will receive 100 mg of modafinil capsules for 1 week, followed by 200 mg for 7 weeks (as long as the drug is well tolerated), which they will take daily in the morning. During this time, participants will complete questionnaires and neurocognitive tests, and report adverse events at study visits.
  Other Names: Provigil; Alertec; 2-benzhydrylsulfinylacetamide
  Arms: Modafinil
Drug: Placebo — Participants randomized to the placebo group will receive 100 mg placebo capsules for 1 week, followed by 200 mg for 7 weeks, which they will take daily in the morning. During this time, participants will complete questionnaires and neurocognitive tests, and report adverse events at study visits.
  Arms: Placebo

SUMMARY:
Cognitive difficulties such as indecisiveness or inability to concentrate are core symptoms of depression with up to 90% of untreated depressed individuals experiencing these symptoms. As many as half of those who remit from a major depressive episode continue to experience residual cognitive deficits, but these symptoms are frequently overlooked in clinical practice. This leads to persistent cognitive deficits which can cause reduced level of functioning and loss of productivity. As standard antidepressants have an inadequate impact on these residual cognitive symptoms, further treatment options are required. Modafinil is a wakefulness agent with evidence that it improves some domains in cognition such as memory in those whose non-cognitive depressive symptoms have been treated over a short term period. This medication may have favourable lasting effects on cognition, such as the ability to plan and execute tasks in those who receive modafinil for a longer time period. The aim of this study is to investigate whether modafinil can enhance cognition and have additional effects on functioning and work productivity in a sample of participants who were treated for depression but who continue to experience cognitive deficits.

DETAILED DESCRIPTION:
Background:

Major Depressive Disorder (MDD) is a chronic mental disorder with a lifetime prevalence of 5-20% (Kessler et al., 2003; Woo et al., 2016). While depressed mood and loss of interest in activities are core features of MDD, cognitive deficits such as indecisiveness and inattention are present and interfere with work and social functioning (McIntyre et al., 2013). These cognitive deficits frequently persist beyond remission from a Major Depressive Episode (MDE), with up to 94% of those impaired during an episode continuing to experience deficits after the episode (Bhalla et al., 2006), including deficits in attention, executive functioning, and psychomotor speed (Salagre et al., 2017). These residual cognitive symptoms often persist and are associated with poor functioning and loss of productivity (Lam et al., 2014).

In a systematic review examining MDD patients in remission, multiple regression analyses found that MDD predicted lower performance on measures of attention, processing speed, and cognitive flexibility relative to healthy controls (HCs; Hasselbalch et al., 2011). Further evidence for the presence of neuropsychological deficits in remitted MDD patients comes from a systematic review and meta-analysis that found the remitted MDD patient group had executive function and attentional deficits, while symptomatic patients exhibited executive function, attentional, and memory deficits (Roc et al., 2013).

Importantly, there are no medications with evidence to modify cognition in remitted depression. This suggests that in order to assist in the recovery of cognitive and functional abilities, additional novel treatment options are required.

There is considerable evidence that subjective and objective measures of cognition are not well correlated in MDD. This has informed the investigators' choice of separate subjective and objective measures for this study. In addition, cognitive disturbances affect psychosocial function and quality of life across several areas, and this necessitated measurement of quality of life. In this study, the investigators will use a computerized version of the Central Nervous System (CNS) Vital Signs Cognitive Battery, which will provide a Neurocognitive Index score (NCI). The NCI is a global measure of cognitive functioning, averaging the scores from 7 tests over 5 domains: composite memory, psychomotor speed, reaction time, complex attention, and cognitive flexibility.

Pilot results from the The Canadian Biomarker Integration Network in Depression (CAN-BIND)-1 study, involving treatment with escitalopram, have clearly documented the nature of deficits, and are in line with expectations in remitted depression. In this pilot sample of 208 participants, 15% of participants had global cognitive impairment despite 8 weeks of antidepressant treatment and achievement of clinical remission (McInerney, personal communication).

In an 8-week antidepressant study, those who significantly improved in global cognitive functioning (assessed using NCI) had superior functioning and work productivity relative to those who did not significantly improve (Hasselbalch et al., 2011). Vortioxetine is the only antidepressant with modest evidence for improving cognitive parameters during a depressive episode (Rock et al., 2013). Research into the use of psychostimulants as a treatment for cognitive deficits in depressed patients has led to the consideration of modafinil and methylphenidate as potential novel pharmacological treatments (Minzenberg et al., 2008). Modafinil is a well-tolerated wakefulness agent where only two clinical studies have previously examined its role on cognition in depression; one where currently depressed patients had improvements in one measure of executive function after 4 weeks of treatment as an adjuvant (DeBattista et al., 2004), and the other where there were improvements in memory after a single dose in depressed participants who achieved remission (Kaser et al., 2016). Unlike methylphenidate, modafinil appears to impact both "hot" (emotion-laden) and "cold" (independent of emotion) cognitive deficits, which are commonly seen in remitted depression.

Immediate effects of modafinil on cognition have been shown (Kaser et al., 2016) and the investigators will be the first to examine the pro-cognitive effects in a remitted depressed sample over 8 weeks. The dose of modafinil (200mg) used in the study, sample size, and randomized control trial (RCT) study design parallels those described in the immediate effect study, and this maintains continuity. However, the study does not examine whether the immediate effects are maintained. More importantly, it is unclear whether the cognitive improvements translate into improvement in functioning.

The added focus on functional outcomes fits with patient-centered models of healthcare, as functional outcomes are of greatest importance to most patients. Thus, the RCT study and choice of outcome variables have been carefully designed with specific endpoints to delineate these aspects. Cognitive flexibility, memory, and attention will be domains of importance in this study, since these domains have been shown in previous literature to be improved by modafinil (Minzenberg et al., 2008; DeBattista et al., 2004; Kaser et al., 2016).

Objectives, Hypotheses, and Impact:

The primary objective of this study is to delineate the cognitive effects of modafinil in patients with remitted depression at baseline and 4 weeks, and monitor whether these effects are maintained with continual dosage over an 8-week period. The secondary objective of this study is to understand the effect of modafinil in patients with remitted depression on measures of functioning at baseline, 4 weeks, and 8 weeks, and whether these effects parallel the cognitive changes.

The investigators' overarching hypothesis is that specific aspects of cognitive functioning, including the domains of memory, attention, and cognitive flexibility, will improve through treatment with modafinil. The investigators hypothesize that participants with remitted depression who continue to experience cognitive deficits and are taking modafinil will have improvements in aspects of cognitive domains at 4 weeks, and these improvements will be sustained at 8 weeks. It is also hypothesized that functional improvements will parallel the improvements in cognitive domains.

The study ensures a closer examination of modafinil's effect on individual facets of cognition in patients with remitted MDD. This enhanced understanding will enable the development of new treatment plans for residual cognitive symptoms, where none currently exist. Moreover, it could spur interest in new drug development programs to address an unmet need of targeting cognition across disorders where depression is a central feature (e.g. Bipolar Disorder, Generalized Anxiety Disorder). Finally, the study would delineate the specific endophenotypes within cognition (e.g. working memory) and functional improvement (e.g. social functioning), which would lead to personalized treatment options based on the endophenotype profile.

Methods In this randomized control trial, remitted MDD patients with residual cognitive deficits (n=50) will have cognitive symptoms and functioning evaluated before and after an 8-week trial of modafinil 200mg or placebo. Participants will be recruited through the ongoing CAN-BIND 1 Wellness Study; the Depression Program at St. Michael's Hospital; the shared care network at St. Michael's Hospital; and referrals from residents, family doctors, and other St. Michael's psychiatrists. All participants who meet inclusion criteria will be asked to enrol in this study and provide written informed consent.

Participants will be on a stable dose of an antidepressant for at least 6 months prior to enrolment. They will be required to remain on this stable dose for the duration (8 weeks) of the trial. They will be prescribed modafinil or placebo at a dose of 100 mg for the first week then 200mg for 7 weeks. After week 8, participants will be informed of which group they were in and if they were taking modafinil, they can choose to continue on modafinil or to discontinue.

Participants will undergo an 8-week randomized, placebo controlled treatment trial of modafinil 200mg with a total of 3 study visits. Participants may require more clinical visits as needed. Screening will be done to confirm study eligibility. At the screening visit all participants will provide demographic data (age, gender, education, ethnicity, occupation, family history of mental illness), undergo a structured diagnostic assessment (Mini-International Neuropsychiatric Interview), complete the CNS Vital Signs cognitive battery, and have the Montgomery-Asberg Depression Rating Scale administered. At the baseline visit, participants will initiate the study drug trial, complete clinician rated and self-report scales, and complete the cognitive battery in CNS Vital Signs. Participants will start with a 100 mg dose at baseline, and increase to the 200 mg dose at week 1 if the drug is well tolerated. Participants will repeat all measures at week 4 and 8. Adverse events will be recorded at each study visit. For participants who wish to discontinue the study drug at week 8, they will first have their dose decreased to 100 mg for one week and attend an additional week 9 safety visit to evaluate adverse events before full discontinuation of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual (DSM)-5 criteria for past Major Depressive Episode within MDD, confirmed through Mini-International Neuropsychiatric Interview (MINI) diagnosis
2. Age between 18 and 55 years
3. Montgomery-Åsberg Depression Rating Scale < 7 (in remission)
4. Ability to read and understand English
5. Participant has been treated with an antidepressant for ≥ 6 months prior to enrolment
6. Participant agrees to remain on a stable antidepressant regimen for the duration of the trial (8 weeks)
7. Participant is currently experiencing cognitive deficits, as confirmed by an NCI >1 standard deviation below the mean on CNS Vital Signs cognitive battery
8. Women of child bearing potential must agree to use birth control for the duration of the study and 1 month following discontinuation of the study drug

Exclusion Criteria:

1. Pregnancy/lactation
2. Lifetime history of Bipolar I, II or psychosis; other comorbidities (e.g. Generalized Anxiety, Panic Disorder) may be allowed by clinician judgement
3. Subject has current clinical diagnosis of autism, dementia, intellectual disability, or mild cognitive impairment
4. Meets DSM-5 criteria for active Post-Traumatic Stress Disorder, confirmed through MINI diagnosis
5. Subject meets criteria for current personality disorder
6. Concomitant use of monoamine oxidase inhibitors and/or other psychotropic drugs including lithium, clomipramine, and triazolam
7. Recent (< 6 months) stimulant use, such as medications used for attention deficit hyperactivity disorder
8. Subject is taking antipsychotics
9. Subject is taking herbaceuticals (i.e. natural products that have psychoactive properties, such as St. John's wort)
10. Concomitant use of medications that may interact with modafinil, including warfarin and cyclosporine
11. Medical condition requiring immediate investigation or treatment
12. Recent (< 6 months)/current history of drug abuse/dependence (other than caffeine or nicotine)
13. Previous intolerance or failure to respond to an adequate trial of modafinil
14. Any past history of head injury or concussion, as confirmed by the Ohio State University Traumatic brain injury (TBI) Identification Short Form
15. Current suicidal ideation (MADRS Item 10 ≤2 or by clinician judgement)
16. History of coronary artery disease, recent (<1 year) myocardial infarction, or unstable angina
17. History of left ventricular hypertrophy, ischemic ECG changes, chest pain, arrhythmia, or clinically significant manifestations of mitral valve prolapse in association with use of CNS stimulants
18. Involvement in another treatment study during the time of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Cognition | 8 weeks
  Cognition will be measured using a Neurocognitive Index, which will be calculated using the CNS Vital Signs Neurocognitive Battery (a computer program). The domains tested within the cognitive battery include composite memory, psychomotor speed, reaction time, complex attention, cognitive flexibility, and processing speed. The Neurocognitive Index is based on a composite, average score of the scores on these 6 domains. From the Neurocognitive Index score, the CNS Vital Signs program classifies the participant as above, average, low average, low, or very low based on their deviation from a standard score of 85.

SECONDARY OUTCOMES:
Composite Memory | 8 weeks
  This is a measure of how well participants can recognize, remember, and retrieve words and images. Composite memory will be measured based on performance on a series of tests in the CNS Vital Signs Neurocognitive Battery (a computer program). Based on performance, the CNS Vital Signs program classifies the participant as above, average, low average, low, or very low based on their deviation from a standard score of 103.
Psychomotor Speed | 8 weeks
  This is a measure of how well a participant is able to perceive, attend, and respond to complex visual-perceptual information and perform simple, fine motor coordination. Psychomotor speed will be measured based on performance on a series of tests in the CNS Vital Signs Neurocognitive Battery (a computer program). Based on performance, the CNS Vital Signs program classifies the participant as above, average, low average, low, or very low based on their deviation from a standard score of 93.
Reaction Time | 8 weeks
  This is a measure of how quickly a participant can react to simple and complex direction sets. Reaction time will be measured based on performance on a series of tests in the CNS Vital Signs Neurocognitive Battery (a computer program). Based on performance, the CNS Vital Signs program classifies the participant as above, average, low average, low, or very low based on their deviation from a standard score of 107.
Complex Attention | 8 weeks
  This is a measure of a participant's ability to track and respond to multiple stimuli over long periods of time, and perform complex mental tasks quickly and accurately. Complex attention will be measured based on performance on a series of tests in the CNS Vital Signs Neurocognitive Battery (a computer program). Based on performance, the CNS Vital Signs program classifies the participant as above, average, low average, low, or very low based on their deviation from a standard score of 56.
Cognitive Flexibility | 8 weeks
  This is a measure of how well a participant can adapt to rapidly changing and complex directions, and manipulate information. Cognitive flexibility will be measured based on performance on a series of tests in the CNS Vital Signs Neurocognitive Battery (a computer program). Based on performance, the CNS Vital Signs program classifies the participant as above, average, low average, low, or very low based on their deviation from a standard score of 63.
Processing Speed | 8 weeks
  This is a measure of a participant's ability to recognize and process information. Processing speed will be measured based on performance on a series of tests in the CNS Vital Signs Neurocognitive Battery (a computer program). Based on performance, the CNS Vital Signs program classifies the participant as above, average, low average, low, or very low based on their deviation from a standard score of 79.
Subjective Cognitive Improvement | 8 weeks
  This is a measure of how well the participant feels their cognition has improved after using the study drug. This will be measured using the British Columbia Cognitive Complaints Inventory, a 6-item screening tool that assesses perceived cognitive difficulties in patients with MDD over the past 7 days. A total score between 0 and 18 is calculated based on participant self-report, where a higher score represents greater cognitive impairment.
Functional Disability | 8 weeks
  This will be assessed using the Sheehan Disability Scale, which assesses functional impairment in work/school, social life, and family life. This is scored based on a self-report scale of 0-10 in 3 domains: work/school, social life, and family life/home responsibilities. A total score between 0 and 30 is calculated based on the sum of these 3 domains. Higher values represent greater disability.
Work Productivity | 8 weeks
  This will be assessed using the Lam Employment and Productivity Scale, a brief questionnaire designed to assess occupational productivity.This is scored based on a self-report scale from 0-4 in 7 domains: low energy or motivation, poor concentration or memory, anxiety or irritability, getting less work done, doing poor quality work, making more mistakes, and having trouble getting along with people or avoiding them. A total score between 0 and 28 is calculated as a sum of all sub scores. Higher values represent greater impairment.
Motivation and Energy | 8 weeks
  This is be assessed using the Motivation and Energy Inventory, an 18-item inventory to measure changes in lassitude and energy with antidepressant treatment. Based on self-report measurements, a total score between 0-108 is determined, where a lower score corresponds to lower levels of motivation and energy.

OTHER OUTCOMES:
Overall Quality of Life | 8 weeks
  This will be assessed using the World Health Organization Quality of Life, Shortened Version. A score between 4 and 20 is determined for four domains: physical health, psychological health, social relationships, and environment. A total score for overall quality of life between 16 and 80 is then calculated as the sum of these four domain scores. A higher score represents greater quality of life.
Life Enjoyment and Satisfaction | 8 weeks
  This is measured using the Quality of Life Enjoyment and Satisfaction Questionnaire, a depression-specific quality of life measure. This questionnaire is scored using 8 domains: physical health/activities (possible score between 13-65), feelings (total score between 14-70), work (total score between 13-65), household duties (total score between 10-50), school/course work (total score between 10-50), leisure time activities (total score between 6-30), social relations (total score between 11-55), and overall satisfaction (total score between 12-60). Lower scores represent lower levels of enjoyment and satisfaction.
Sleepiness | 8 weeks
  This will be assessed using the Epworth Sleepiness Scale, an 8-item scale used as a subjective measure of a patient's sleepiness. A total score between 0 and 24 is calculated based on the participant's self-report, where higher scores represent greater sleepiness.
Fatigue | 8 weeks
  This will be assessed using the Fatigue Severity Scale, a 9-item questionnaire with questions related to how fatigue interferes with certain activities. A total score between 9 and 63 is calculated based on the participant's self-report, where higher scores represent greater levels of fatigue.
Sleep Quality | 8 weeks
  This will be assessed using the Pittsburgh Sleep Quality Index, which assesses night-time sleep problems, focusing on sleep experiences over the past month. A total score between 0 and 21 is assigned, where higher scores represent worse sleep quality.
Depressive Symptomatology | 8 weeks
  This will be assessed using 2 measures. The first is the Quick Inventory of Depressive Symptomatology, a 6-item measure of MDD symptom severity; a total score between 0-27 is possible for this questionnaire based on participant self-report. The second measure is the Montgomery-Asberg Depression rating scale, a clinician-administered 10-item scale that incorporates symptoms most sensitive to change; a total score of 0-60 is possible. Both of these scores will be converted to percentages (i.e. participant score divided by total possible score) and then averaged to get a final percentage representing depressive symptoms. A higher score represents a higher degree of depressive symptoms.
Anxiety Symptomatology | 8 weeks
  Th is measured using the Generalized Anxiety Disorder 7-Item, an anxiety scale used for assessing anxiety severity. A total score is calculated based on 7 questions (each of which are self-rated on a scale of 0 to 3) for a total score between 0 and 21. Higher scores represents a higher degree of anxiety symptoms.
Psychiatric Symptomatology | 8 weeks
  This will be assessed using the Brief Symptom Inventory-53, which assesses the psychological profile of an individual covering somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. A global severity index is determined as the mean score on the 53 questions on this inventory. Each question is self-rated by the participant on a scale of 0 to 4, and a total score of 0 to 4 is possible for the global severity index. A higher score represents a higher degree of psychiatric symptoms.
Treatment Satisfaction (with study drug) | 8 weeks
  This will be assessed by administering the Abbreviated Treatment Satisfaction Questionnaire for Medication, a 9-item questionnaire evaluating patient satisfaction with medication treatment in a study. A total score of 9 to 59 is possible, where higher scores represent greater treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sidney H Kennedy, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Woo YS, Rosenblat JD, Kakar R, Bahk WM, McIntyre RS. Cognitive Deficits as a Mediator of Poor Occupational Function in Remitted Major Depressive Disorder Patients. Clin Psychopharmacol Neurosci. 2016 Feb 29;14(1):1-16. doi: 10.9758/cpn.2016.14.1.1. PMID 26792035
- [Background] McIntyre RS, Cha DS, Soczynska JK, Woldeyohannes HO, Gallaugher LA, Kudlow P, Alsuwaidan M, Baskaran A. Cognitive deficits and functional outcomes in major depressive disorder: determinants, substrates, and treatment interventions. Depress Anxiety. 2013 Jun;30(6):515-27. doi: 10.1002/da.22063. Epub 2013 Mar 6. PMID 23468126
- [Background] Bhalla RK, Butters MA, Mulsant BH, Begley AE, Zmuda MD, Schoderbek B, Pollock BG, Reynolds CF 3rd, Becker JT. Persistence of neuropsychologic deficits in the remitted state of late-life depression. Am J Geriatr Psychiatry. 2006 May;14(5):419-27. doi: 10.1097/01.JGP.0000203130.45421.69. PMID 16670246
- [Background] Salagre E, Sole B, Tomioka Y, Fernandes BS, Hidalgo-Mazzei D, Garriga M, Jimenez E, Sanchez-Moreno J, Vieta E, Grande I. Treatment of neurocognitive symptoms in unipolar depression: A systematic review and future perspectives. J Affect Disord. 2017 Oct 15;221:205-221. doi: 10.1016/j.jad.2017.06.034. Epub 2017 Jun 19. PMID 28651185
- [Background] Lam RW, Kennedy SH, Mclntyre RS, Khullar A. Cognitive dysfunction in major depressive disorder: effects on psychosocial functioning and implications for treatment. Can J Psychiatry. 2014 Dec;59(12):649-54. doi: 10.1177/070674371405901206. No abstract available. PMID 25702365
- [Background] Hasselbalch BJ, Knorr U, Kessing LV. Cognitive impairment in the remitted state of unipolar depressive disorder: a systematic review. J Affect Disord. 2011 Nov;134(1-3):20-31. doi: 10.1016/j.jad.2010.11.011. Epub 2010 Dec 15. PMID 21163534
- [Background] Rock PL, Roiser JP, Riedel WJ, Blackwell AD. Cognitive impairment in depression: a systematic review and meta-analysis. Psychol Med. 2014 Jul;44(10):2029-40. doi: 10.1017/S0033291713002535. Epub 2013 Oct 29. PMID 24168753
- [Background] Minzenberg MJ, Carter CS. Modafinil: a review of neurochemical actions and effects on cognition. Neuropsychopharmacology. 2008 Jun;33(7):1477-502. doi: 10.1038/sj.npp.1301534. Epub 2007 Aug 22. PMID 17712350
- [Background] DeBattista C, Lembke A, Solvason HB, Ghebremichael R, Poirier J. A prospective trial of modafinil as an adjunctive treatment of major depression. J Clin Psychopharmacol. 2004 Feb;24(1):87-90. doi: 10.1097/01.jcp.0000104910.75206.b9. PMID 14709953
- [Background] Kaser M, Deakin JB, Michael A, Zapata C, Bansal R, Ryan D, Cormack F, Rowe JB, Sahakian BJ. Modafinil Improves Episodic Memory and Working Memory Cognition in Patients With Remitted Depression: A Double-Blind, Randomized, Placebo-Controlled Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2017 Mar;2(2):115-122. doi: 10.1016/j.bpsc.2016.11.009. PMID 28299368